CLINICAL TRIAL: NCT00474929
Title: A Phase I/II Study of the Raf Kinase/VEGFR Inhibitor Sorafenib in Combination With the mTOR Inhibitor RAD001 (Everolimus) in Patients With Relapsed Non-Hodgkin Lymphoma, Hodgkin Lymphoma, or Multiple Myeloma
Brief Title: Sorafenib and Everolimus in Treating Patients With Relapsed or Refractory Lymphoma or Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LS0689; 07-000710 (Other: Mayo Clinic IRB); LS0689 (Other: Mayo Clinic Cancer Center ID)
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Results first posted 2016-07-07 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-02

CONDITIONS: Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm
Keywords: recurrent adult Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage III multiple myeloma; refractory multiple myeloma; Waldenström macroglobulinemia; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; cutaneous B-cell non-Hodgkin lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent adult grade III lymphomatoid granulomatosis
MeSH Terms: conditions — Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Waldenstrom Macroglobulinemia; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Mycosis Fungoides; Sezary Syndrome | interventions — Everolimus; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multiple Myeloma (Experimental): Phase I: Dose level 0: Sorafenib 200 mg twice daily, RAD001 5mg every other day; Dose level 1: Sorafenib 200 mg twice daily, RAD001 5mg every day; Dose level 2: Sorafenib 400 mg twice daily, RAD001 5mg every day; Dose level 3: Sorafenib 400 mg twice daily, RAD001 10mg every day; Phase II: Sorafenib 200 mg twice daily, RAD001 5mg every day;
  Interventions: Drug: RAD001; Drug: Sorafenib
- Lymphoma (Experimental): Phase I: Dose level 0: Sorafenib 200 mg twice daily, RAD001 5mg every other day; Dose level 1: Sorafenib 200 mg twice daily, RAD001 5mg every day; Dose level 2: Sorafenib 400 mg twice daily, RAD001 5mg every day; Dose level 3: Sorafenib 400 mg twice daily, RAD001 10mg every day; Phase II: Sorafenib 200 mg twice daily, RAD001 5mg every day;
  Interventions: Drug: RAD001; Drug: Sorafenib

INTERVENTIONS:
Drug: RAD001 — Phase I: Dose level 0: RAD001 5mg every other day; Dose level 1: RAD001 5mg every day; Dose level 2: RAD001 5mg every day; Dose level 3: RAD001 10mg every day; Phase II: RAD001 5mg every day;
  Other Names: Everolimus
Drug: Sorafenib — Phase I: Dose level 0: Sorafenib 200 mg twice daily; Dose level 1: Sorafenib 200 mg twice daily; Dose level 2: Sorafenib 400 mg twice daily; Dose level 3: Sorafenib 400 mg twice daily; Phase II: Sorafenib 200 mg twice daily;
  Other Names: sorafenib tosylate

SUMMARY:
RATIONALE: Sorafenib and everolimus may stop the growth of cancer cells by blocking blood flow to the cancer and by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I/II trial is studying the side effects and best dose of sorafenib and everolimus and to see how well they work in treating patients with relapsed or refractory non-Hodgkin's lymphoma, Hodgkin's lymphoma, or multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose (MTD) of sorafenib tosylate and everolimus in patients with relapsed or refractory non-Hodgkin's lymphoma, Hodgkin's lymphoma, or multiple myeloma.
* Determine the toxicity of this regimen in these patients.
* Evaluate the therapeutic activity of this regimen in these patients.
* Evaluate the pharmacokinetic interaction of this regimen.
* Correlate clinical (toxicity and/or tumor response or activity) effects with pharmacologic (pharmacokinetic/pharmacodynamic) parameters and/or biologic (correlative laboratory) results.

OUTLINE: This is a multicenter, dose-escalation, phase I study followed by a phase II study.

* Phase I (closed to accrual as of 2/10/2009): Patients receive oral sorafenib tosylate and oral everolimus on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of sorafenib tosylate and everolimus until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 out of at most 6 patients experience a Dose Limiting Toxicity (DLT).

* Phase II: Patients receive oral sorafenib tosylate twice daily and oral everolimus once daily at the MTD determined in phase I. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Blood and bone marrow are collected periodically during the study and analyzed by flow cytometry, immunohistochemistry, and enzyme-linked immunosorbent assay. Patients enrolled in phase I also undergo blood sample collection on days 8 and 15 during course 1 and on day 1 of each subsequent course for pharmacokinetic studies.

After completion of study treatment, patients are followed every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 103 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed diagnosis of 1 of the following:

  * Multiple myeloma
  * Non-Hodgkin's lymphoma
  * Hodgkin's lymphoma
* Relapsed or refractory disease
* Measurable disease, as defined according to diagnosis as follows:

  * Multiple myeloma, meeting 1 of the following criteria:

    * Serum monoclonal protein ≥ 1.0 g/dL
    * Urine monoclonal protein ≥ 200 mg by 24-hour electrophoresis
    * Serum immunoglobulin free light chain ≥ 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
    * Monoclonal bone marrow plasmacytosis ≥ 30% (evaluable disease)
  * Lymphoma, meeting 1 of the following criteria:

    * Measurable disease by CT scan or MRI or PET/CT scan, defined as ≥ 1 lesion that has a single diameter of ≥ 2 cm OR tumor cells in the blood ≥ 5 x10^9/L

      * Skin lesions can be used if the area is ≥ 2 cm in ≥ 1 diameter and photographed with a ruler
  * Lymphoplasmacytic lymphoma without measurable lymphadenopathy, meeting both of the following criteria:

    * Bone marrow lymphoplasmacytosis with > 10% lymphoplasmacytic cells or aggregates, sheets, lymphocytes, plasma cells, or lymphoplasmacytic cells on bone marrow biopsy
    * Quantitative IgM monoclonal protein > 1,000 mg/dL
* Not a candidate for known standard potentially curative therapy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* ANC ≥ 1,500/mm³
* Hemoglobin ≥ 9 g/dL
* Platelet count ≥ 75,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN) OR direct bilirubin normal
* AST ≤ 3 times ULN (5 times ULN if liver involvement)
* Creatinine ≤ 2.5 times ULN
* INR < 1.5 or activated PTT < 1.5 times ULN (no concurrent anticoagulants)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for at least 2 weeks after completion of study treatment
* No uncontrolled infection
* No NYHA class III-IV congestive heart failure
* No unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months)
* No myocardial infarction within the past 6 months
* No uncontrolled hypertension, defined as systolic blood pressure (BP) > 150 mm Hg or diastolic BP > 90 mm Hg, despite optimal medical management
* No known HIV positivity
* No other active malignancy requiring treatment
* No inability to swallow
* No gastrointestinal (GI) function impairment or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative disease, uncontrolled nausea, vomiting, or diarrhea, malabsorption syndrome, or small bowel resection) or preclude use of oral medications
* No thrombolic or embolic events (e.g., cerebrovascular accident, including transient ischemic attacks) within the past 6 months
* No pulmonary hemorrhage or bleeding event ≥ grade 3 within the past 4 weeks
* No severe or uncontrolled medical conditions or other conditions that would preclude study compliance
* No liver disease, such as cirrhosis, chronic hepatitis or chronic persistent hepatitis, or uncontrolled infections
* No serious nonhealing wound, ulcer, or bone fracture
* No evidence or history of serious bleeding diathesis or coagulopathy, such as hemophilia or von Willebrand's disease
* No significant traumatic injury within the past 4 weeks
* No known hypersensitivity to everolimus or other rapamycins (sirolimus, temsirolimus)

PRIOR CONCURRENT THERAPY:

* More than 3 weeks since prior myelosuppressive chemotherapy or biological therapy and recovered
* More than 4 weeks since prior major surgery or open biopsy

  * Lymph node biopsy within past 4 weeks allowed
* Prior everolimus allowed
* No concurrent immunosuppressant therapy

  * Concurrent stable chronic doses of steroids (≤ 20 mg of prednisone per day) for disorders other than lymphoma (i.e., rheumatoid arthritis, polymyalgia rheumatica, adrenal insufficiency, asthma) or for pruritus or fever associated with lymphoma allowed
  * Concurrent corticosteroids at the lowest possible dose necessary to control symptoms in patients with CNS lymphoma allowed
* No concurrent CYP450 enzyme-inducing antiepileptic drugs (e.g., phenytoin, carbamazepine, or phenobarbital), rifampin, or Hypericum perforatum (St. John's wort)
* No other concurrent immunotherapy, radiotherapy, or chemotherapy
* No concurrent chronic oxygen therapy
* No concurrent warfarin or heparin
* No other concurrent investigational therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2007-08-29 (Actual); Primary Completion 2011-11-05 (Actual); Study Completion 2019-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Witzig, MD, Principal Investigator — Mayo Clinic; Shaji K. Kumar, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Mayo Clinic Cancer Center, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I, Dose Level 0: Phase I: Dose level 0: Sorafenib 200 mg twice daily, RAD001 5mg every other day
- Phase I, Dose Level 1: Phase I: Dose level 1: Sorafenib 200 mg twice daily, RAD001 5mg every day
- Phase I, Dose Level 2: Phase I: Dose level 2: Sorafenib 400 mg twice daily, RAD001 5mg every day
- Phase I, Dose Level 3: Phase I: Dose level 3: Sorafenib 400 mg twice daily, RAD001 10mg every day
- Phase II: Phase II: Sorafenib 200 mg twice daily, RAD001 5mg every day;
Period: Overall Study
Arm/Group | Phase I, Dose Level 0 | Phase I, Dose Level 1 | Phase I, Dose Level 2 | Phase I, Dose Level 3 | Phase II
Started | 6 | 6 | 7 | 7 | 77
Completed | 6 | 5 | 5 | 5 | 77
Not Completed | 0 | 1 | 2 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Not completed — Unrelated medical condition | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I, Dose Level 0: Phase I: Dose level 0: Sorafenib 200 mg twice daily, RAD001 5mg every other day;
- Total: Total of all reporting groups
Arm/Group | Phase I, Dose Level 0 | Phase I, Dose Level 1 | Phase I, Dose Level 2 | Phase I, Dose Level 3 | Phase II | Total
Number analyzed (Participants) | 6 | 5 | 5 | 5 | 77 | 98
Age, Continuous [Median (Full Range); unit: years] | 43 [22 to 64] | 63 [50 to 67] | 56 [43 to 63] | 61 [24 to 69] | 61 [22 to 83] | 61 [22 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 1 | 30 | 36
  Male | 3 | 4 | 4 | 4 | 47 | 62
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 5 | 5 | 77 | 98

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting a Dose Limiting Toxicity (DLT)
Description: The Maximum Tolerated Dose (MTD) is defined as the dose level below the lowest dose that induces dose-limiting toxicity (DLT) in at least one-third of patients (at least 2 of a maximum of 6 new patients). Dose-limiting toxicity (DLT) is defined as an adverse event attributed (definitely, probably, or possibly) in first cycle to the study treatment and meeting the following criteria:
  * Grade 4 infection
  * Grade 4 ANC or PLT
  * Grade 3 or higher non-hematologic adverse event.
  NCI Common Terminology Criteria for Adverse Events (CTCAE) v3.0 will be used to assess adverse events. For this endpoint, the number of patients reporting a DLT event are tabulated.
Time Frame: First cycle (28 days) of study treatment
Measure: Number; unit: participants
Groups:
- Phase I, Dose Level 1: Dose level 1: Sorafenib 200 mg twice daily, RAD001 5mg every day
- Phase I, Dose Level 2: Dose level 2: Sorafenib 400 mg twice daily, RAD001 5mg every day
- Phase I, Dose Level 3: Dose level 3: Sorafenib 400 mg twice daily, RAD001 10mg every day
Arm/Group | Phase I, Dose Level 0 | Phase I, Dose Level 1 | Phase I, Dose Level 2 | Phase I, Dose Level 3
Number analyzed (Participants) | 6 | 5 | 5 | 5
participants | 1 | 0 | 1 | 2
Statistical Analysis 1: Comparison: Phase I, Dose Level 0 vs Phase I, Dose Level 1 vs Phase I, Dose Level 2 vs Phase I, Dose Level 3; The Maximum Tolerated Dose (MTD) is defined as the dose level below the lowest dose that induces dose-limiting toxicity (DLT) in at least one-third of patients (at least 2 of a maximum of 6 new patients); Test type: Superiority or Other; Maximum Tolerated Dose (MTD) Level = 1 — Dose Level 1 was chosen as the MTD due to PI concerns about adverse events and frequent dose reductions seen on later cycles at dose level 2. For the best interest of the patients, dose level 1 was chosen as the MTD and the dose level for Phase II

2. Primary Outcome: Proportion of Confirmed Tumor Responses
Description: A confirmed response is defined to be a CR or PR noted as the objective status for eligible patients during cycles 1-12.
  Complete Response (CR):
  * Multiple Myeloma (MM): Negative immunofixation of serum and urine, disappearance of soft tissue plasmacytomas, and normalization of free light chain (FLC) ratio.
  * Lymphoma: Disappearance of all clinical and radiographic evidence of disease, all lymph nodes of normal size (1.5 cm or less), no splenomegaly.
  Partial Response (PR):
  * MM: 50% reduction of serum or urine M-protein or to less than 200mg/day, a 50% reduction in the difference between involved and uninvolved FLC, and 50% reduction in the size of soft tissue plasmacytoma.
  * Lymphoma: 50% or greater reduction in sum of the products of the dimension for nodal masses; no increase in liver, spleen or node size; no new sites of disease; and a 50% decrease in lymphocyte count if followed at baseline.
Time Frame: Up to 12 cycles of treatment
Measure: Number; unit: percentage of participants
Groups:
- Sorafenib 200 mg Twice Daily, RAD001 5mg Every Day: This endpoint was analyzed using all patients treated at the MTD (Dose Level 1: Sorafenib 200 mg twice daily, RAD001 5mg every day). Due to concerns about adverse events and frequent dose reductions seen on later cycles at dose level 2, the PI felt it was in the best interest of the patients to choose dose level 1 as the MTD and the dose level for Phase II.
  Therefore, the analysis of the Phase II endpoint includes the eligible Phase I participants treated at Dose Level 1 (N=5) and it includes all participants treated in Phase II (N=77).
Arm/Group | Sorafenib 200 mg Twice Daily, RAD001 5mg Every Day
Number analyzed (Participants) | 82
percentage of participants
  Complete Response (CR) | 8.5
  Partial Response (PR) | 15.9

3. Secondary Outcome: Survival Time
Description: Survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 3 years from registration
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Sorafenib 200 mg Twice Daily, RAD001 5mg Every Day: This endpoint was analyzed using all patients treated at the MTD (Dose Level 1: Sorafenib 200 mg twice daily, RAD001 5mg every day). This includes the eligible Phase I participants treated at Dose Level 1 (N=5) and it includes all participants treated in Phase II (N=77).
Arm/Group | Sorafenib 200 mg Twice Daily, RAD001 5mg Every Day
Number analyzed (Participants) | 82
months | 13.5 [10.3 to 21.1]

4. Secondary Outcome: Progression Free Survival
Description: Progression Free Survival is defined as the time from registration to the earliest date documentation of disease progression or death. The distribution of time to disease progression will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 3 years from registration
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib 200 mg Twice Daily, RAD001 5mg Every Day
Number analyzed (Participants) | 82
months | 4.6 [3.6 to 6.2]

ADVERSE EVENTS:
Time Frame: The adverse events reported here occurred during treatment. The maximum treatment length was 27, 28-day cycles.
Description: Adverse events were collected at the end of each cycle.
Arm/Group | Phase I, Dose Level 0 | Phase I, Dose Level 1 | Phase I, Dose Level 2 | Phase I, Dose Level 3 | Phase II
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/5 | 2/5 | 1/5 | 22/77
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5 | 5/5 | 5/5 | 76/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I, Dose Level 0 (N=6) | Phase I, Dose Level 1 (N=5) | Phase I, Dose Level 2 (N=5) | Phase I, Dose Level 3 (N=5) | Phase II (N=77)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infectious colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Platelet count decreased (Investigations) | 1 (2) | 1 (1) | 1 (1) | 1 (2) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I, Dose Level 0 (N=6) | Phase I, Dose Level 1 (N=5) | Phase I, Dose Level 2 (N=5) | Phase I, Dose Level 3 (N=5) | Phase II (N=77)
Hemoglobin decreased (Blood and lymphatic system disorders) | 3 (13) | 2 (2) | 4 (12) | 3 (15) | 31 (63)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (12) | 2 (8) | 3 (10) | 5 (20) | 53 (266)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (3) | 16 (35)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (7) | 2 (4) | 3 (6) | 4 (5) | 35 (90)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (7) | 1 (2) | 1 (3) | 4 (6) | 20 (27)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (6)
Fatigue (General disorders) | 6 (33) | 4 (7) | 4 (19) | 4 (26) | 67 (357)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (3)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (7)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intraoperative respiratory injury - Nasal cavity (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7)
Alkaline phosphatase increased (Investigations) | 1 (3) | 1 (3) | 1 (1) | 0 (0) | 4 (12)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 4 (4)
Laboratory test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukocyte count decreased (Investigations) | 2 (6) | 1 (1) | 1 (1) | 5 (18) | 23 (50)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 6 (23)
Neutrophil count decreased (Investigations) | 2 (2) | 2 (5) | 1 (1) | 5 (20) | 19 (34)
Platelet count decreased (Investigations) | 3 (8) | 2 (4) | 2 (5) | 3 (22) | 32 (99)
Serum cholesterol increased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Weight loss (Investigations) | 1 (1) | 1 (1) | 1 (4) | 0 (0) | 2 (6)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 6 (8)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (8)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 1 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (7) | 1 (2) | 3 (8) | 2 (2) | 10 (27)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum triglycerides increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (8)
Taste alteration (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (6) | 2 (13) | 16 (78)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 4 (10) | 0 (0) | 3 (4) | 5 (8) | 42 (105)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (7) | 1 (1) | 1 (3) | 1 (4) | 18 (76)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes